CLINICAL TRIAL: NCT02743923
Title: Chemotherapy in KRAS Mutated Chemotherapy Naive Non-small Cell Lung Cancer Patients: a Phase III Study Comparing Cisplatin-pemetrexed With Carboplatin-paclitaxel-bevacizumab: NVALT 22
Brief Title: Cisplatin-Pemetrexed Compared With Carboplatin-Paclitaxel-Bevacizumab in KRAS Mutated Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVALT 22
Record Dates: First submitted 2016-03-17; First posted 2016-04-19 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Bevacizumab; Pemetrexed; Cisplatin

ARMS (2):
- carboplatin-paclitaxel- bevacizumab (Active Comparator): carboplatin AUC 6, paclitaxel 200 mg/m2, bevacizumab 15 mg/kg all administered intravenously on day 1 every 3 weeks for 4-6 cycles, followed by bevacizumab maintenance every 3 weeks until progression
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: Bevacizumab
- cisplatin-pemetrexed (Active Comparator): pemetrexed 500 mg/m2 administered intravenously on day 1 and cisplatin 75 mg/m2 administered intravenously on day 1 every 3 weeks for 4-6 cycles, followed by maintenance pemetrexed every 3 weeks until progression.
  Interventions: Drug: Pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: carboplatin — AUC 6
  Arms: carboplatin-paclitaxel- bevacizumab
Drug: paclitaxel — 200mg/m2
  Arms: carboplatin-paclitaxel- bevacizumab
Drug: Bevacizumab — 15 mg/kg
  Arms: carboplatin-paclitaxel- bevacizumab
Drug: Pemetrexed — 500 mg/m2
  Arms: cisplatin-pemetrexed
Drug: cisplatin — 75 mg/m2
  Arms: cisplatin-pemetrexed

SUMMARY:
The purpose of this study is to determine whether carboplatin-paclitaxel-bevacizumab results in a prolonged progression free survival compared to cisplatin-pemetrexed as first line treatment in patients with KRAS mutated non-small cell lung cancer.

DETAILED DESCRIPTION:
KRAS mutations occur in 30% of patients with non-small cell lung cancer, especially adenocarcinoma. For long time KRAS mutation has been related with poor prognosis and poor response to chemotherapy. Recent data however show that this is both not true. It seems that response, progression free survival and overall survival is similar in KRAS mutated. Until now no specific targeted therapy is available for KRAS mutated NSCLC patients. Optimization of treatment in advanced NSCLC patients with a KRAS mutation could also be achieved by selecting the best available chemotherapy treatment.

Two standard chemotherapy schemes are frequently used and FDA and EMA approved as first line treatment for patients with adenocarcinoma: cisplatin-pemetrexed and carboplatin-paclitaxel-bevacizumab.

The aim of this randomized phase III study is to compare two standard treatment regimens in patients with KRAS mutated, advanced stage NSCLC and the hypothesis is that bevacizumab with chemotherapy improves outcomes compared to chemotherapy alone as first line treatment. Furthermore the outcome for the different KRAS mutations will be studied.

Treatment with one of the two following chemotherapy combinations according to the label: carboplatin-paclitaxel-bevacizumab or cisplatin-pemetrexed q3wks for up to six cycles. Continuation maintenance with bevacizumab and pemetrexed is allowed until progression. Blood and archival tissue will be optionally collected for translational research. This may help to identify subgroups of patients who are likely better treated with a specific treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed (non-squamous) NSCLC incurable locally advanced or metastatic (stage IIIB and stage IV) disease.
2. Documented KRAS mutation
3. Chemotherapy-naive NSCLC patients. Adjuvant chemotherapy or chemoradiotherapy is allowed when given > 1 year for study entry. Previous anti-PD(L1) therapy for advanced disease is allowed.
4. At least one unidimensionally measurable lesion meeting RECIST1.1.
5. ECOG PS 0-2
6. Age ≥ 18 years
7. Adequate organ function, including:

   * Adequate bone marrow reserve: ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L.
   * Hepatic: bilirubin ≤1.5 x ULN, AP, ALT, AST ≤ 3.0 x ULN AP, ALT, and AST ≤5 xULN is acceptable if the liver has tumor involvement
   * Renal: calculated creatinine clearance ≥ 60 ml/min based on the Cockroft-Gault formula.
   * Urine protein (dip-stick) < 2 +; when ≥ 2 +: 24 hours urine protein ≤ 1 gr.
8. Signed informed consent
9. Male and female patients with reproductive potential must use an approved contraceptive method, if appropriate. Female patients with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

1. Pregnant or lactating women
2. Clinically significant (i.e. active) cardiovascular disease: congestive heart failure >NYHA class 2; CVA or myocardial infarction < 6 months prior to study entry; uncontrolled hypertension (blood pressure systolic > 150 mmHg and/or diastolic > 100 mmHg)
3. History of hemoptysis ≥ grade 2 (bright red blood of at least 2,5 ml in the last 3 months)
4. Evidence of tumor invading major blood vessels on imaging (i.e. superior vena cava or pulmonary artery)
5. Patients with evidence or history of bleeding diathesis
6. Non-healing wound or ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
progression free survival | Every 6 weeks, from date of randomization until the date of progression of disease or of death from any cause, assessed up to 60 months

SECONDARY OUTCOMES:
disease control rate | Every 6 weeks, from date of randomization until the date of progression of disease or of death from any cause, assessed up to 60 months.
overall survival | date of randomization to the date of death from any cause, assessed up to 60 months.
  Stratification for KRAS mutation (G12V versus G12C versus other)
outcome between G12V versus G12C versus other subtypes of KRAS mutations (mutational analysis on plasma and blood platelets). | date of randomization to the date of death from any cause, assessed up to 60 months.
  The two most common KRAS types are G12C in about 40% of cases, G12V in 18% and G12D in 15% of cases. Subgroup analyses are planned to explore treatment effect in these different KRAS mutations groups. At baseline the metastatic patterns of these subgroups will be described. KRAS mutations in NSCLC occur mainly in codon 12 and 13.
  Stratification for KRAS mutation (G12V versus G12C versus other) at randomization.
response by Crabb criteria (if applicable) | Every 6 weeks, from date of randomization until the date of progression of disease or of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie C Dingemans, MD PhD, Principal Investigator — Dutch Society of Physicians for Pulmonology and Tuberculosis
Locations (28):
- Netherlands (28):
  - VUmc Medical Center, Amsterdam, North Holland
  - Medical spectrum Twente, Enschede, Overijssel
  - Meander Medical Center, Amersfoort, Utrecht
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - ZGT, Almelo
  - Antoni van Leeuwenhoek, Amsterdam
  - OLVG, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Amphia Hospital, Breda
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Maxima Medisch Centrum, Eindhoven
  - Groene Hart, Gouda
  - UMCG, Groningen
  - Martini Ziekenhuis, Groningen
  - Tergooi ziekenhuizen, Hilversum
  - Spaarne Gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maastricht University Medical Center, Maastricht
  - Maasstad ziekenhuis, Rotterdam
  - St. Fransicus Gasthuis, Rotterdam
  - Haga, The Hague
  - Medical Center Haaglanden, The Hague
  - Diakonessenhuis Utrecht, Utrecht
  - St. Antonius ziekenhuis, Utrecht
  - VieCuri Medisch Centrum voor Noord-Limburg, Venlo
  - Isala Klinieken, Zwolle